CLINICAL TRIAL: NCT02399007
Title: A Prospective, Randomized, Multicenter, Controlled Study Comparing the Outcomes of Primary Total Hip Arthroplasty Devices Manufactured in China Versus Devices Manufactured Outside of China
Brief Title: A Clinical Trial Study of Hip System in Primary Total Hip Arthroplasty in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Medical (Suzhou) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPS-201301
Record Dates: First submitted 2015-03-20; First posted 2015-03-26 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Rheumatoid Arthritis; Congenital Hip Dysplasia; Avascular Necrosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Hip Dislocation, Congenital; Osteonecrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Hip System made in China (Experimental): Patient in this arm will be implanted with Primary Total Hip Arthroplasty Devices Manufactured in China
  Interventions: Device: Total Hip System made in China (SUN, CoCr, Duraloc, Marathon)
- Total Hip System made outside of China (Active Comparator): Patient in this arm will be implanted with Primary Total Hip Arthroplasty Devices Manufactured Outside of China
  Interventions: Device: Total Hip System made outside of China (Summit, CoCr, Duraloc, Marathon)

INTERVENTIONS:
Device: Total Hip System made in China (SUN, CoCr, Duraloc, Marathon) — SUN Hip stem,CoCr Femoral Head,Duraloc Porocoat Sector acetabular shell,Marathon 10D polyethylene liner (ETO)
  Arms: Total Hip System made in China
Device: Total Hip System made outside of China (Summit, CoCr, Duraloc, Marathon) — Summit Porocoat STD,CoCr Femoral Head,Duraloc Porocoat Sector acetabular shell,Marathon 10D polyethylene liner (ETO)
  Arms: Total Hip System made outside of China

SUMMARY:
A clinical trial of total Hip system used in Primary Total Hip Arthroplasty in China.

DETAILED DESCRIPTION:
A Prospective, Randomized, Multicenter, Controlled Study Comparing the Outcomes of Primary Total Hip Arthroplasty Devices Manufactured in China versus Devices Manufactured Outside of China

ELIGIBILITY:
Inclusion Criteria:

1. The subject is ≥55, and ≤80 years old
2. The Subject must be of Chinese ethnic descent and be willing to return on three occasions for clinical evaluations.
3. Subject is a suitable candidate for primary total hip replacement using the devices described in this CIP
4. Subject must meet all criteria specified in BOTH SUN hip stem and Summit hip stem instructions for use (IFU)
5. Before surgery, subject is willing and able to sign the informed consent form approved by the Institutional Review Board (IRB), Ethics Committee (EC) or Ethical Review Board (ERB).
6. Subject, in the opinion of the Clinical Investigator, is able to understand this clinical investigation and co-operate with investigational procedures.
7. Subject must be comfortable with speaking, reading, and understanding questions and providing responses in an available translated language for the patient reported outcomes (PROs) in the CIP.
8. Subject is receiving a unilateral hip replacement or, if a contralateral hip replacement is anticipated, the surgery must occur within 6 months of the first study hip. The second hip will not be enrolled in the study.

Exclusion Criteria:

1. Subject does not provide written voluntary consent to participate in the clinical study.
2. The Subject is a woman who is pregnant or lactating.
3. Subjects who have undergone THA in contralateral hip within the past 6 months.
4. Contralateral hip has been enrolled in the study.
5. Presence of any previous prosthetic hip replacement device in affected hip.
6. Previous Girdlestone procedure (resection arthroplasty) or surgical fusion of the affected hip
7. Subject has hip dysplasia CROWE classification grade of 3 or 4.
8. Above knee amputation of either contralateral or ipsilateral leg
9. Subject is anticipated to require a contralateral THA between 6 months and 1-year.
10. Subject has an active infection
11. Subject has a malignant disease, severe condition, alcohol or drug addiction and/or mental disorders that the investigator believes will interfere with the study participation.
12. Subjects with severe osteoporosis, metabolic bone disease, radioactive bone disease or tumor in the bone surrounding the hip joint that, in the opinion of the investigator, will negatively impact implant fixation and the outcome of the investigation;
13. Subject has significant neurological or musculoskeletal disorders or disease that may adversely affect gait or weight bearing (e.g. muscular dystrophy, multiple sclerosis, cerebral infarction, hemiplegia, Charcot disease).
14. Subject is not comfortable with speaking, reading, and understanding questions and providing responses in an available translated language for the PROs in the CIP.
15. Subject has a medical condition with less than 2 years of life expectancy due to other medical conditions.
16. The patient has comorbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study.
17. The patient is currently participating in another investigational drug or device study.
18. Subject is a prisoner.
19. Subject has a known allergy to any component of the implant (metal for example).

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-06-07 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Harris Hip Total Score at 12 months postoperatively | 12 months postoperatively

SECONDARY OUTCOMES:
One year non-revision rate where revision is defined as removal of any component for any reason with the exception of infection | 12 months postoperatively
One year non-revision rate where revision is defined as removal of any component secondary to infection | 12 months postoperatively

OTHER OUTCOMES:
Harris Hip Total Score success: success is ≥ 80 points. | 12 months postoperatively
Patient Reported Outcomes | Preoperation to 12 months postoperatively
  SF 12: scores at 1 yr, change from pre-op. WOMAC: scores at 1 yr., change from pre-op.
Radiographs: incidence of clinically relevant radiolucent lines, and osteolysis | Preoperation to 12 months postoperatively
Adverse Events: tally the type and frequency of adverse events | Preoperation to 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Shigui Yan, Principal Investigator — The second Affiliated Hospital of Zhejiang Medicine University
Locations (8):
- China (8):
  - The first affiliated hospital of Guangzhou Tranditional Meidical University, Guangzhou, Guangdong
  - The third affiliated hospital of Hebei University, Shijiazhuang, Hebei
  - The second affiiliated hospital of Harbin Medical University, Harbin, Heilongjiang
  - The first affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - The affiliated hosoital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xinjiang Medicine University, Hohhot, Xinjiang
  - The general hospital of Kunming, Kunming, Yunnan
  - The second Affiliated Hospital of Zhejiang Medicine University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No